CLINICAL TRIAL: NCT05392023
Title: Effects of Scapular Stabilization Program on Pain, Range of Motion and Disability in Patients With Chronic Non- Specific Neck Pain
Brief Title: Effects of Scapular Stabilization Program in Patients Chronic Non-specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0143 Moeen
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Neck Pain
Keywords: Neck pain; Scapular stabilization program; Neck Disability Index
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Scapular Stabilization exercise program
  Interventions: Other: Relaxation Exercises and Scapular Stabilization exercise program
- Group B (Other): Relaxation Exercises of cervico- scapular region
  Interventions: Other: Relaxation Exercises of cervico- scapular region

INTERVENTIONS:
Other: Relaxation Exercises and Scapular Stabilization exercise program — Scapular Stabilization Program (3 sets of 10 reps each/day). This exercise program is for muscles affecting scapular alignment due to chronic neck pain. A specialized program of non-resistive scapular upward rotation, wall facing arm lift, backward rolling arm lift, overhead arm raise, shoulder abduction in scapular plane above 120˚, shoulder shrugs, levator scapulae and pectoralis minor stretching. Hot pack (10 min) and relaxation exercises including myofascial release and stretching of neck and scapular region muscles. A total of 45 minutes session three times a week on alternate days for 3 weeks. Assessment will be done at baseline, on the end of 3rd week and for long-term effects at the end of 6th week.
  Arms: Group A
Other: Relaxation Exercises of cervico- scapular region — Relaxation exercises of the cervico-scapular region including neck stretches of scapular muscles and myofascial release will be given to patients three times a week on alternate days for 3 weeks. Assessment will be done at baseline, at the end of the 3rd week, and for long-term effects at the end of the 6th week.
  Arms: Group B

SUMMARY:
The aim of this study is to determine the effects of scapular stabilization program on pain, range of motion and disability in patients with chronic non- specific neck pain. This study will be a randomized controlled trial and 28 patients fulfilling the inclusion criteria will be included in the study. they will be allocated into 2 groups using non- probability purposive sampling technique. Experimental group will receive relaxation exercises for the cervico-scapular region combined with SSP(scapular stabilization program). The Control group will receive relaxation exercises only. Outcome measure: Numeric Pain Rating Scale, Goniometer, and Neck Disability Index will measure pain, range of motion, and disability. The experimental group will receive a total of 45 minutes sessions, thrice a week on alternate days for 3 weeks. The Control group will receive relaxation exercises in cervico-scapular region including neck stretches, stretches of scapular muscles, and myofascial release 3 times a week for 3 weeks on alternate days. Measurements will be taken at the baseline, at the end of 3rd week and for long term effects follow- up at 6 weeks. Data will be analyzed by SPSS version 20.

DETAILED DESCRIPTION:
This study will provide evidence for management strategies of chronic NNP (nonspecific neck pain) solely focusing on a well-designed SSP (scapular stabilization program). The study will enable physiotherapists to induct this exercise program (Scapular stabilization program) in their treatment regimens to manage NNP. Some studies have used these exercises in combination to treat people with chronic neck pain. It is hypothesized that adding a scapular stabilization program will increase treatment efficacy. This study will enable us to solely evaluate the effects of SSP on NNP without adding other treatment strategies. This study aims to determine the effects of a scapular stabilization program on pain, range of motion and disability in patients with chronic non-specific neck pain. This study will be a randomized controlled trial and 28 patients fulfilling the inclusion criteria will be included in the study. they will be allocated into 2 groups using the non-probability purposive sampling technique. The experimental group will receive relaxation exercises for the cervico-scapular region combined with SSP(scapular stabilization program). The Control group will receive relaxation exercises only. Outcome measure: Numeric Pain Rating Scale, Goniometer and Neck Disability Index will measure pain, range of motion, and disability. The experimental group will receive a total of 45 minutes sessions, thrice a week on alternate days for 3 weeks. The Control group will receive relaxation exercises in the cervico-scapular region including neck stretches, stretches of scapular muscles, and myofascial release 3 times a week for 3 weeks on alternate days. Measurements will be taken at the baseline, at the end of the 3rd week and for long-term effects follow up at the 6th week. Data will be analyzed by SPSS version 20.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age between 18-35 years

  * NPRS value more than or equal to 4
  * Chronic nonspecific neck pain for more than 3 months
  * Shoulder flexion 130˚ or more

Exclusion Criteria:

* Structural abnormalities like fractures/spondylosis

  * Any other musculoskeletal problem
  * Neurological problems
  * H/o cervical or thoracic surgery Psychological disorders

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 3rd day
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10) that best reflects the intensity of his/her pain 11-point numeric scale ranges from '0' representing no pain to 10 representing the worst imaginable pain
Goniometer | 3rd day
  The science of measuring the joint ranges in each plane of the joint is called goniometry. Goniometer is a device that measures an angle or permits the rotation of an object to a definite position. Thoracic flexion and extension will be assessed through it.
NDI | 3rd day
  It is a 10-item questionnaire that measures a patient's self-reported neck pain related disability.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil-ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Melo Castro Deligne L, Rocha MCB, Malta DC, Naghavi M, de Azeredo Passos VM. The burden of neck pain in Brazil: estimates from the global burden of disease study 2019. BMC Musculoskelet Disord. 2021 Sep 21;22(1):811. doi: 10.1186/s12891-021-04675-x. PMID 34548044
- [Background] Sadeghian F, Raei M, Amiri M. Persistent of Neck/Shoulder Pain among Computer Office Workers with Specific Attention to Pain Expectation, Somatization Tendency, and Beliefs. Int J Prev Med. 2014 Sep;5(9):1169-77. PMID 25317301
- [Background] Mahmud N, Bahari SF, Zainudin NF. Psychosocial and ergonomics risk factors related to neck, shoulder and back complaints among Malaysia office workers. International Journal of Social Science and Humanity. 2014;4(4):260-3.
- [Background] Haldeman S, Carroll L, Cassidy JD. Findings from the bone and joint decade 2000 to 2010 task force on neck pain and its associated disorders. J Occup Environ Med. 2010 Apr;52(4):424-7. doi: 10.1097/JOM.0b013e3181d44f3b. PMID 20357682
- [Background] Helgadottir H, Kristjansson E, Mottram S, Karduna AR, Jonsson H Jr. Altered scapular orientation during arm elevation in patients with insidious onset neck pain and whiplash-associated disorder. J Orthop Sports Phys Ther. 2010 Dec;40(12):784-91. doi: 10.2519/jospt.2010.3405. Epub 2010 Oct 22. PMID 20972341
- [Background] Yildiz TI, Turgut E, Duzgun I. Neck and Scapula-Focused Exercise Training on Patients With Nonspecific Neck Pain: A Randomized Controlled Trial. J Sport Rehabil. 2018 Sep 1;27(5):403-412. doi: 10.1123/jsr.2017-0024. Epub 2018 Jul 25. PMID 28605288
- [Background] Cagnie B, Struyf F, Cools A, Castelein B, Danneels L, O'leary S. The relevance of scapular dysfunction in neck pain: a brief commentary. J Orthop Sports Phys Ther. 2014 Jun;44(6):435-9. doi: 10.2519/jospt.2014.5038. Epub 2014 May 10. PMID 24816504
- [Background] Sihawong R, Janwantanakul P, Sitthipornvorakul E, Pensri P. Exercise therapy for office workers with nonspecific neck pain: a systematic review. J Manipulative Physiol Ther. 2011 Jan;34(1):62-71. doi: 10.1016/j.jmpt.2010.11.005. PMID 21237409
- [Background] Andersen CH, Andersen LL, Zebis MK, Sjogaard G. Effect of scapular function training on chronic pain in the neck/shoulder region: a randomized controlled trial. J Occup Rehabil. 2014 Jun;24(2):316-24. doi: 10.1007/s10926-013-9441-1. PMID 23832167
- [Background] Kang JI, Choi HH, Jeong DK, Choi H, Moon YJ, Park JS. Effect of scapular stabilization exercise on neck alignment and muscle activity in patients with forward head posture. J Phys Ther Sci. 2018 Jun;30(6):804-808. doi: 10.1589/jpts.30.804. Epub 2018 Jun 12. PMID 29950768